CLINICAL TRIAL: NCT04567628
Title: The Relationship Between Vedolizumab Therapeutic Drug Monitoring, Biomarkers of Inflammation and Clinical Outcomes in the Real World Setting (VEDO TDM RWE)
Brief Title: Study of Relationship Between Vedolizumab Therapeutic Drug Monitoring, Biomarkers of Inflammation and Clinical Outcomes
Acronym: VEDO TDM RWE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-5062; U1111-1256-3663 (Registry Identifier: WHO)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TDM Cohort: Participants diagnosed with inflammatory bowel disease (IBD) (UC or CD) within Takeda Canada Patient Support Program (PSP) group who received treatment with vedolizumab 300 milligram (mg), infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and TDM at pre-specified intervals during their treatment were observed retrospectively.
  Interventions: Other: No Intervention
- Historical Cohort: Participants diagnosed with IBD (UC or CD) within Takeda Canada PSP group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 but did not undergo biomarker testing or TDM during their treatment were observed retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — As this was an observational study, no intervention was administered.

SUMMARY:
The purpose of this study is to determine if a relationship exists between Week 6 vedolizumab therapeutic drug monitoring (TDM) and Week 30 Faecal calprotectin (FCP).

DETAILED DESCRIPTION:
This is a non-interventional, retrospective, and longitudinal study of participants with IBD (UC or CD) receiving vedolizumab between years 2015 and 2020. The study will determine the real-world evidence of vedolizumab, its relationship with TDM, biomarkers of inflammation, and its effect on clinical outcomes in a real-world setting.

This study will enroll approximately 5,500 participants. Participants will be enrolled in 2 cohorts: TDM Cohort and Historical Cohort. The study will have a retrospective data collection of the participants from PSP between the years 2015 and 2020. The study will include longitudinal analysis of data collected in a subset of Takeda Canada PSP, specifically for those participants on vedolizumab, some of which received biomarker testing and TDM at pre-specified intervals during their treatment.

This multi-center trial will be conducted in Canada. The overall time for data collection in the study will be approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or, when applicable, the participant's legally acceptable representative signed and dated a written, informed consent form, which specified secondary use of their data, and any required privacy authorization as part of their enrollment in Takeda Canada's PSP.
2. Received or receiving vedolizumab between the years 2015 and 2020.

Exclusion Criteria:

No exclusion criteria will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with IBD (UC or CD) receiving vedolizumab between years 2015 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 7873 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Takeda Canada, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Seow CH, Marshall JK, Stewart E, Pettengell C, Ward R, Afif W. The relationship among vedolizumab drug concentrations, biomarkers of inflammation, and clinical outcomes in a Canadian real-world study. J Can Assoc Gastroenterol. 2024 Mar 24;7(4):290-298. doi: 10.1093/jcag/gwae010. eCollection 2024 Aug. PMID 39139218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Canada from 05 October 2020 to 22 September 2021.
Pre-assignment Details: Data of participants diagnosed with moderate to severe inflammatory bowel disease (IBD)- Crohn's disease (CD) or ulcerative colitis (UC) was analyzed retrospectively in this observational study. Total of 7873 participants entered the patient support program, out of which 5194 participants met study criteria, had non-missing therapeutic drug monitoring (TDM) Week 6 values, and were analyzed.
Groups:
- TDM Cohort: Participants diagnosed with IBD (UC or CD) within Takeda Canada Patient Support Program (PSP) group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and therapeutic drug monitoring (TDM) at pre-specified intervals during their treatment were observed retrospectively.
Period: Overall Study
Arm/Group | TDM Cohort | Historical Cohort
Started | 436 | 4758
Completed | 436 | 4758
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analyzed participants included all participants who were not screen failures, met all the inclusion criteria and had enough information about response to the biological treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | TDM Cohort | Historical Cohort | Total
Number analyzed (Participants) | 436 | 4758 | 5194
Age, Customized [Count of Participants; unit: Participants]
  Less Than 18 Years | 0 | 0 | 0
  18 Years and Above | 436 | 4758 | 5194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 2370 | 2591
  Male | 215 | 2388 | 2603
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 436 | 4758 | 5194

OUTCOME MEASURES:

1. Primary Outcome: TDM Cohort: Correlation Between Week 6 Vedolizumab TDM and Week 30 Faecal Calprotectin (FCP)
Description: The relationship between vedolizumab TDM at Week 6 and FCP levels at Week 30 were studied using univariate and multivariate logistic regression models. Multivariate analyses were performed to control for possible confounding factors such as age, sex, disease type (CD/UC), duration, prior immunomodulator/biologic therapy, vedolizumab start and end dates, vedolizumab dose, vedolizumab frequency, and albumin. FCP was used as a surrogate marker for disease severity, and by extension drug efficacy. The FCP level was detected in participant's stool 30 weeks after the participant's first dose of vedolizumab. FCP was treated as a continuous variable for correlation analysis to determine Spearman's correlation coefficient. This outcome measure was planned to be analyzed only in participants enrolled in the TDM Cohort.
Time Frame: After the first dose of vedolizumab (at Week 30)
Population: as for baseline characteristics
Measure: Number; unit: correlation coefficient
Groups:
- TDM Cohort: Participants diagnosed with IBD (UC or CD) within Takeda Canada PSP group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and TDM at pre-specified intervals during their treatment were observed retrospectively. FCP was treated as a continuous variable for correlation analysis to determine Spearman's correlation coefficient. This outcome measure was planned to be analyzed only in participants enrolled in the TDM Cohort.
Arm/Group | TDM Cohort
Number analyzed (Participants) | 436
correlation coefficient | -0.23
Statistical Analysis 1: Comparison: TDM Cohort; Test type: Other; p = 0.003, Spearman's Rank Correlation

2. Secondary Outcome: TDM Cohort: C-reactive Protein (CRP) Level at Week 30
Description: The CRP level were detected in participant's blood 30 weeks after the participant's first dose of vedolizumab. CRP was used as a surrogate marker for disease severity, and by extension drug efficacy. This outcome measure was planned to be analyzed separately in participants with UC and CD who were collectively a part of the TDM Cohort.
Time Frame: After the first dose of vedolizumab (at Week 30)
Population: Analyzed participants included all participants who were not screen failures, met all the inclusion criteria and had enough information about response to the biological treatment. Overall number analyzed are the number of participants with data available for analyses.
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- TDM Cohort: Ulcerative Colitis: Participants diagnosed with IBD (UC) within Takeda Canada PSP group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and TDM at pre-specified intervals during their treatment were observed retrospectively.
- TDM Cohort: Crohn's Disease: Participants diagnosed with IBD (CD) within Takeda Canada PSP group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and TDM at pre-specified intervals during their treatment were observed retrospectively.
Arm/Group | TDM Cohort: Ulcerative Colitis | TDM Cohort: Crohn's Disease
Number analyzed (Participants) | 91 | 119
mg/L | 2 [1 to 5] | 3 [1 to 6]
Statistical Analysis 1: Comparison: TDM Cohort: Ulcerative Colitis vs TDM Cohort: Crohn's Disease; Test type: Other; p = 0.25, Log Rank — A two-sided p-value of <0.05 was considered statistically significant

3. Secondary Outcome: TDM Cohort: Disease Score for Crohn's Disease (CD) Participants Based on Harvey-Bradshaw Index (HBI) at Week 30
Description: Disease activity scores of CD participants were based on HBI. It consists of clinical parameters: general well-being (0 = very well to 4 = terrible), abdominal pain (0 = none to 3 = severe), number of liquid or soft stools per day, abdominal mass (0 = none to 3 = definite and tender), and complications (8 items; 1 score per item). The total score is sum of sub scores, where score <5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and >16 = severe disease activity. This outcome measure was planned to be analyzed only in participants with CD.
Time Frame: After the first dose of vedolizumab (at Week 30)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TDM Cohort: Crohn's Disease
Number analyzed (Participants) | 67
score on a scale | 3 [1 to 6]

4. Secondary Outcome: TDM Cohort: Disease Score for Ulcerative Colitis (UC) Participants Based on Partial Mayo Score at Week 30
Description: Disease activity scores of UC participants were based on Partial Mayo score. It consists of 3 sub-scores: stool pattern, most severe rectal bleeding of the day, and global assessment by physician, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9. Here, higher scores indicate more severe disease. This outcome measure was planned to be analyzed only in participants with UC.
Time Frame: After the first dose of vedolizumab (at Week 30)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | TDM Cohort: Ulcerative Colitis
Number analyzed (Participants) | 46
score on a scale | 1 [0 to 3]

5. Secondary Outcome: Number of Participants Categorized Based on Dose Escalation
Description: Dose escalation was defined as a change from doses every 8 weeks to every 4 weeks.
Time Frame: Baseline (Week 0) up to Week 30 (after first dose of vedolizumab)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- TDM Cohort: Participants diagnosed with IBD (UC or CD) within Takeda Canada PSP group who received treatment with vedolizumab 300 mg, infusion, intravenously, at Weeks 0, 2, and 6, and every 8 weeks thereafter as per product Health Canada Product Monograph, or every 4 or 6 weeks thereafter as per standard clinical practice between the year 2015 to 2020 along with the biomarker testing and TDM at pre-specified intervals during their treatment were observed retrospectively.
Arm/Group | TDM Cohort | Historical Cohort
Number analyzed (Participants) | 436 | 4758
Participants | 173 | 852
Statistical Analysis 1: Comparison: TDM Cohort vs Historical Cohort; Test type: Other; p < 0.001, Log Rank — A two-sided p-value of <0.05 was considered statistically significant

6. Secondary Outcome: TDM Cohort: Number of Participants Categorized Based on Treatment Persistence at the End of the TDM Study at Week 30
Description: Treatment persistence was defined as whether the participant was still on the treatment at the end of the TDM study. This outcome measure was planned to be analyzed only in participants enrolled in the TDM Cohort.
Time Frame: After the first dose of vedolizumab (at Week 30)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | TDM Cohort
Number analyzed (Participants) | 436
Participants
  Treatment Persistence | 360
  Did not Persist on Treatment | 76

7. Secondary Outcome: Treatment Duration
Description: Treatment duration was defined as the length of time a participant remains on treatment (i.e., from the year 2015 to 2020).
Time Frame: From treatment initiation up to discontinuation of treatment or up to data extraction date Oct 2020), whichever occurs first (maximum up to approximately 5 years)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TDM Cohort | Historical Cohort
Number analyzed (Participants) | 436 | 4758
days | 378.0 [238.0 to 553.5] | 242.0 [116.0 to 437.5]
Statistical Analysis 1: Comparison: TDM Cohort vs Historical Cohort; Test type: Other; p < 0.0001, Log Rank — A two-sided p-value of <0.05 was considered statistically significant

ADVERSE EVENTS:
Time Frame: From enrollment on 5 October 2020 to last date of assessment 22 September 2021 (Up to approximately 12 months)
Description: As Adverse Events (serious and non-serious) were not part of the study objectives and endpoints, data was not abstracted or collected from healthcare records or other applicable source records.
Arm/Group | TDM Cohort | Historical Cohort
All-Cause Mortality (participants affected / at risk) | 0/436 | 0/4758
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04567628/Prot_SAP_000.pdf